CLINICAL TRIAL: NCT05407909
Title: To Evaluate the Safety and Tolerability of SYHX2001 in Patients With Advanced or Metastatic Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: CSPC ZhongQi Pharmaceutical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SYHX2001C101
Record Dates: First submitted 2022-05-30; First posted 2022-06-07 (Actual); Last update posted 2022-08-09 (Actual); Status verified 2022-08

CONDITIONS: Advanced or Metastatic Solid Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SYHX2001 (Experimental): SYHX2001 will be administered orally.
  Interventions: Drug: SYHX2001

INTERVENTIONS:
Drug: SYHX2001 — SYHX2001 tablets, oral

SUMMARY:
This is a Phase 1, open-label, multicenter, dose escalation and expansion study to evaluate the safety, tolerability, pharmacokinetics, and pharmacodynamics of the experimental drug(SYHX2001) in previously treated patients with advanced or metastatic cancer.

DETAILED DESCRIPTION:
This is a multicenter, open-label, dose-escalation, dose-expansion Phase 1 study of SYHX2001(name of the experimental drug) in patients with advanced or metastatic cancers who have exhausted standard treatment. The study will consist of 2 parts, a dose escalation part and a cohort expansion part. Once the recommended phase 2 dose (RP2D) has been determined in the dose escalation part, a cohort expansion part involving up to three separate cohorts will be conducted. For patients, the study will include a screening phase, a treatment phase, and a post treatment follow-up phase. An end-of-study visit will be conducted within 30 days after the last dose of SYHX2001.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients with an age of 18~75years (inclusive).
2. Confirmed histologic or cytologic diagnosis of an advanced and/or metastatic solid tumor.
3. At least one measurable lesion as defined by RECIST version 1.1.
4. Eastern Cooperative Oncology Group Performance Status 0 or 1.
5. Life expectancy ≥3 months.
6. Major organ function within 14 days prior to treatment meets the following criteria (no blood transfusion, Erythropoietin(EPO), Granulocyte Colony Stimulating Factor(G-CSF) or other medical support): Absolute Neutrophil Count(ANC)≥1.5×10^9/L，Platelet(PLT)≥90×10^9/L，Hemoglobin(Hb)≥100g/L or≥6.2 mmol/L；Creatinine(Cr)≤1.5×upper limit of normal(ULN) and creatinine clearance rate≥50mL/min；Total Bilirubin(TBIL)≤1.5×ULN; Prothrombin time(PT)≤1.5×ULN , Activated Partial Thromboplastin Time(APTT)≤1.5×ULN , Aspartate Aminotransferase(AST)/Alanine Aminotransferase(ALT)≤2.5 × ULN.
7. Signed informed consent form.

Exclusion Criteria:

1. Chemotherapy, radiotherapy, biotherapy, endocrine therapy, targeted therapy, immunotherapy and other anti-tumor treatment within 4 weeks prior to the first dose of the study drug, or administration of other investigational agents within 4 weeks or 5 half-lives prior to the first dose of the study drug, whichever is longer.
2. Major surgery or significant trauma within 4 weeks prior to the first dose of the study drug.
3. Adverse reactions from the previous anti-tumor treatment have not yet recovered to ≤ level 1 based on CTCAE 5.0。
4. Have a history of severe cardiovascular and cerebrovascular disease.
5. Central nervous system metastasis or meningeal metastasis with clinical symptoms, or other evidence shows that the patient's central nervous system metastasis or meningeal metastasis has not been controlled and not suitable for the study according to the judgment of the investigator.
6. Known history of hypersensitivity to test drug components.
7. Patients with recent active bleeding or a history of bleeding.
8. Those with coagulation disorders or taking thrombolytic, anticoagulant or antiplatelet agglutination drugs.
9. Gastrointestinal perforation, abdominal fistula, or intra-abdominal abscess within 6 months prior to first dose; or currently under investigator's judgement there are high risk factors for hollow organ perforation/fistula formation).
10. Inability to swallow the drug orally, or a condition that seriously affects gastrointestinal absorption in the judgment of the investigator.
11. Irritable bowel syndrome with signs/symptoms requiring medication.
12. Persistent active diarrhea requiring medical treatment.
13. Concomitant use of strong CYP3A4 inhibitors or inducers, strong CYP2D6 inhibitors and strong P-gp inhibitors within 14 days prior to the first dose of the study drug.
14. History of autoimmune diseases, immunodeficiency, including HIV positive, or other acquired, congenital immunodeficiency, or organ transplant history.
15. Known Hepatitis B Virus (HBV), Hepatitis C Virus (HCV), or other active viral infection.
16. Male and female patients of childbearing potential do not agree to use suitable method of contraception during the treatment and 6 months after the last dose of study medication; female patients do not have negative results of serum/urine pregnancy test within 7 days prior to enrollment and would be breastfeeding.
17. Not suitable for this study as determined by the investigator due to other reasons.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Estimated)
Dates: Start 2022-07-27 (Actual); Primary Completion 2026-01-06 (Estimated); Study Completion 2026-01-06 (Estimated)

PRIMARY OUTCOMES:
Dose limiting toxicities (DLT) in stage Ⅰ | Baseline through Day 28
Maximum tolerated dose (MTD) in stage Ⅰ | Baseline through Day 28
Recommended phase 2 dose (RP2D) | Baseline through approximately 2 years
Incidence and severity of adverse events in stage Ⅰ | Baseline through approximately 2 years
Overall response rate (ORR) in stage Ⅱ | Up to approximately 2 years

SECONDARY OUTCOMES:
Maximum observed plasma concentration (Cmax) of SYHX2001 | Baseline and up to approximately 2 years
Area under the plasma concentration-time curve (AUC) extrapolated from time zero to infinity (AUC[0-inf]) of SYHX2001 | up to approximately 2 years
AUC from time zero to the last quantifiable concentration after dosing (AUC[0-t]) of SYHX2001 | up to approximately 2 years
Terminal phase half-life (t1/2) of SYHX2001 | up to approximately 2 years
Oral clearance (CL/F) of SYHX2001 | up to approximately 2 years
PFS Progression-free survival (PFS) | up to approximately 2 years
  PFS is defined as the time from first dose until radiographic progression per standard criteria or death due to any cause, whichever is earlier.
Duration of Response (DOR) | up to approximately 2 years
  DOR is defined as the time from first evidence of response (complete response or partial response per RECIST 1.1) to earlier date of disease progression or death due to any cause.
Number of patients with any adverse events(AEs) and serious adverse events(SAEs) in stage Ⅱ | up to approximately 2 years
Change from Baseline in symmetrical arginine dimethylation (SDMA) as a pharmacodynamics(PD) measure | Baseline and up to approximately 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Harbin Medical University Cancer Hospital, Harbin, Heilongjiang, China

IPD SHARING:
Plan to Share IPD: Undecided